CLINICAL TRIAL: NCT01385436
Title: Pre-vaccination Distribution of Human Papillomavirus (HPV) Genotypes in Patients With High Grade Cervical Squamous Intraepithelial Lesion (HSIL) and Cervical Cancer From Croatia
Brief Title: Distribution of Human Papillomavirus (HPV) Genotypes in Patients With Cervical Cancer From Croatia
Acronym: HPV-cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital for Infectious Diseases, Croatia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Prof Adriana Vince, MD, PhD, University Hospital for Infectious Diseases, Croatia
Other Study IDs: UHID-02
Record Dates: First submitted 2011-06-24; First posted 2011-06-30 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Cervical Cancer
Keywords: human papillomavirus (HPV); cervical cancer; high grade cervical squamous intraepithelial lesion (HSIL)
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA isolates from biopsy specimens of cervical lesions.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HPV HSIL cervical carcinoma

SUMMARY:
Human papillomavirus (HPV) of high-risk genotype is a necessary risk factor in development of cervical cancer. There is a vaccine available to prevent cervical lesions associated with high-risk HPV genotypes 16 and 18. In Croatia HPV vaccination has not yet been introduced in obligatory vaccination schedule. The aim of this study is to describe the pre-vaccination distribution of HPV genotypes in women with high grade cervical squamous intraepithelial lesion (HSIL) and cervical cancer in Croatia. The investigators hypothesis is that HPV-16 is the most frequently found genotype but the distribution of other HPV genotypes is heterogeneous and includes genotypes currently not covered by vaccination.

DETAILED DESCRIPTION:
This is a single-center cross-sectional study on the molecular virology of human papillomavirus (HPV) in Croatia. The study will enroll women aged 18-65 years of age with cervical intraepithelial neoplasia (CIN2+)cervical lesions that received clinical care at the Croatian Center for Pre-malignant and Malignant Diseases of the Cervix. Women with abnormal cytology (high grade cervical squamous intraepithelial lesion-HSIL, cervical cancer) in the period from 2010 to 2012 will be included. Relevant epidemiological and clinical data will be collected. Biological samples will include both biopsy specimens from cervix and cervical swab. Biological samples will be put in Digene Specimen Transport Medium (Qiagen, Gaithersburg, MD) and further analyzed at the Department of Molecular Diagnostics at the University Hospital for Infectious Diseases in Zagreb. HPV genotyping will be performed by using a standardized molecular assay INNO-LiPA HPV Genotyping Extra Test (Solvay S.A., Brussels, Belgium). Analysis of genomic variants of HPV 16 genotype will be performed by population-based sequencing of L1 genome region.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-65 with a cytological diagnosis of CIN2+cervical lesions from all over Croatia that are referred to National Reference Center because of HSIL or malignant cytology findings

Exclusion Criteria:

* Women younger than 18 or older than 65
* Pregnant women

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 18-65 with a cytological diagnosis of CIN2+cervical lesions from all over Croatia that are referred to the National Reference Center because of HSIL or malignant cytology findings.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Pre-vaccination distribution of HPV genotypes in women with HSIL and invasive cervical carcinoma | two years
  To assess the distribution of different high-risk HPV genotypes in biopsy specimens of 400 women with cytological diagnosis of HSIL and cervical cancer. Biopsy will be performed during colposcopy as a part of of routine clinical work-up in women with abnormal PAP smear finding.

SECONDARY OUTCOMES:
HPV vaccine coverage in Croatia | two years
  To evaluate the percentage of HSIL and cervical cancer that can be prevented by current HPV vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Vince, MD, PhD, Principal Investigator — University Hospital for Infectious Diseases Zagreb, Croatia
Locations (1):
- University Hospital for Infectious Diseases, Croatia, Zagreb, Croatia

REFERENCES:
- [Background] Milutin Gasperov N, Sabol I, Matovina M, Spaventi S, Grce M. Detection and typing of human papillomaviruses combining different methods: polymerase chain reaction, restriction fragment length polymorphism, line probe assay and sequencing. Pathol Oncol Res. 2008 Dec;14(4):355-63. doi: 10.1007/s12253-008-9084-2. Epub 2008 Aug 28. PMID 18752054
- [Background] Lepej SZ, Grgic I, Poljak M, Iscic-Bes J, Skerk V, Vince DB, Dusek D, Vince A. Detection of human papillomavirus genotypes 16/18/45 by hybrid capture hybridisation genotyping probe in clinical specimens: the first report. J Clin Virol. 2007 Oct;40(2):171-2. doi: 10.1016/j.jcv.2007.07.002. Epub 2007 Aug 16. No abstract available. PMID 17702646
- [Background] Seme K, Lepej SZ, Lunar MM, Iscic-Bes J, Planinic A, Kocjan BJ, Vince A, Poljak M. Digene HPV Genotyping RH Test RUO: comparative evaluation with INNO-LiPA HPV Genotyping Extra Test for detection of 18 high-risk and probable high-risk human papillomavirus genotypes. J Clin Virol. 2009 Oct;46(2):176-9. doi: 10.1016/j.jcv.2009.07.017. Epub 2009 Aug 15. PMID 19683958
- [Background] Vrtacnik Bokal E, Kocjan BJ, Poljak M, Bogovac Z, Jancar N. Genomic variants of human papillomavirus genotypes 16, 18, and 33 in women with cervical cancer in Slovenia. J Obstet Gynaecol Res. 2010 Dec;36(6):1204-13. doi: 10.1111/j.1447-0756.2010.01316.x. PMID 21114573
- [Background] Poljak M, Kocjan BJ. Commercially available assays for multiplex detection of alpha human papillomaviruses. Expert Rev Anti Infect Ther. 2010 Oct;8(10):1139-62. doi: 10.1586/eri.10.104. PMID 20954880